CLINICAL TRIAL: NCT02528474
Title: Comparison of Optical Coherence Tomographic Findings After Balloon Angioplasty With Two Different Paclitaxel-Coated Balloons for the Treatment of In-Stent Restenosis in Drug-Eluting Stents
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: As it is difficult to recruit any more subjects, the investigators decided to terminate the study.
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1-2015-0041
Record Dates: First submitted 2015-07-31; First posted 2015-08-19 (Estimated); Last update posted 2019-03-29 (Actual); Status verified 2019-02

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease | interventions — Angioplasty, Balloon

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pantera Lux (Experimental)
  Interventions: Device: balloon angioplasty with Pantera Lux
- SeQuent Please (Active Comparator)
  Interventions: Device: balloon angioplasty with SeQuent Please

INTERVENTIONS:
Device: balloon angioplasty with Pantera Lux — Patient will be considered to be enrolled if ISR in DES was found by angiography. After randomization, patients will be treated with Pantera Lux for treatment of ISR. OCT will be performed just after balloon angioplasty for ISR lesion. Information will be collected and recorded on the treated study vessel including angiographic and OCT parameters. Follow-up OCT at 9 month will be performed.
  Arms: Pantera Lux
Device: balloon angioplasty with SeQuent Please — Patient will be considered to be enrolled if ISR in DES was found by angiography. After randomization, patients will be treated with SeQuent Please for treatment of ISR. OCT will be performed just after balloon angioplasty for ISR lesion. Information will be collected and recorded on the treated study vessel including angiographic and OCT parameters. Follow-up OCT at 9 month will be performed.
  Arms: SeQuent Please

SUMMARY:
Drug-coated balloon technology (DCB) has recently attracted considerable interest as a promising alternative treatment option, particularly in the setting of in-stent restenosis (ISR). Optical coherence tomographic finding of restenosis lesions in drug-eluting stents (DESs) after Balloon Angioplasty with Two Different Paclitaxel-Coated Balloons will be compared between two paclitaxel-coated balloon devices; Pantera Lux™ and SeQuent® Please.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 19 years old
* Patients eligible for percutaneous coronary intervention
* Single or more lesion(s) of restenosis requiring angioplasty in drug-eluting stent
* Reference vessel diameter of target lesion ≥2.5 mm

Exclusion Criteria:

* Cardiogenic shock
* Bifurcation lesion or totally occluded lesion
* Unprotected left main trunk lesion
* Allergies or hypersensitivities to antiplatelet, anticoagulation therapy, contrast media, or paclitaxel
* Heavy calcified (definite calcified lesions on angiogram) or extremely tortuous lesions
* Pregnant women or women with potential childbearing
* Inability to follow the patient over the period of 1 year after enrollment, as assessed by the investigator
* Inability to understand or read the informed content

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2015-09-30; Primary Completion 2017-04-20 (Actual); Study Completion 2017-04-20 (Actual)

PRIMARY OUTCOMES:
Neointimal thickness & area | 9 months
  measured by OCT analysis

CONTACTS AND LOCATIONS:
Locations (1):
- Division of Cardiology, Department of Internal Medicine, Yonsei University College of Medicine, Seoul, South Korea